CLINICAL TRIAL: NCT00401336
Title: Quantification of Liver Iron Overload and Steatosis Using a New Magnetic Resonance Imaging Multiecho Gradient-echo Sequence
Brief Title: Quantification of Liver Iron Overload and Steatosis Using Magnetic Resonance Imaging
Acronym: SURFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGS 2006/0197; PHRC/04-08; CIC0203/044
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Iron Overload; Metabolic Syndrome X; Hepatitis B; Hepatitis C; Alcohol Abuse
Keywords: Magnetic resonance imaging; Hepatic iron; Steatosis
MeSH Terms: conditions — Iron Overload; Metabolic Syndrome; Hepatitis B; Hepatitis C; Alcoholism; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic Resonance Imaging (Experimental): New magnetic resonance imaging multiecho gradient-echo sequence
  Interventions: Device: Magnetic resonance imaging multiecho gradient-echo sequence

INTERVENTIONS:
Device: Magnetic resonance imaging multiecho gradient-echo sequence — Breath-hold gradient echo sequences with a single echo and a new multiple-echo gradient-echo sequence

SUMMARY:
Iron excess is increasingly regarded as an important cofactor in the morbidity attributed to many disorders. Assessment of body iron stores by measurement of serum ferritin concentrations has poor specificity and the most reliable method is histological or biochemical assessment from a liver biopsy. Because liver biopsy is an invasive procedure, imaging methods have been developed to detect and quantify hepatic iron content. The aim of the study is to use a simplified magnetic resonance imaging (MRI) technique to quantify simultaneously iron and fat contents in the liver and to compare the results to the quantification obtained biochemically.

DETAILED DESCRIPTION:
Iron excess is increasingly regarded as an important cofactor in the morbidity attributed to many disorders. Assessment of body iron stores by measurement of serum ferritin concentrations has poor specificity and the most reliable method is histological or biochemical assessment from a liver biopsy. Because liver biopsy is an invasive procedure, imaging methods have been developed to detect and quantify hepatic iron content.

The aim of the study is to use a simplified magnetic resonance imaging technique to quantify simultaneously iron and fat contents in the liver and to compare the results to the quantification obtained biochemically.

Patients who need a liver biopsy will be proposed to be enrolled in the study. A magnetic resonance (MR) study will be performed using breath-hold gradient echo sequences with a single echo and a new multiple-echo gradient-echo sequence. Liver and muscle MR signal will be quantitatively determined and compared to biochemical assessment of liver iron concentration and steatosis quantification.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18,
* Planned liver biopsy (or liver biopsy within 2 months before inclusion) for one of these indications: suspicion of liver iron overload, metabolic syndrome, hepatitis B or C, alcohol abuse. No change in diet, transfusions or iron depletion must have occur between the liver biopsy and the MRI.
* Having given a written informed consent.

Exclusion Criteria:

* Non cooperating patient,
* Patient with dyspnea,
* Patient with contra-indication to MR imaging (pace-maker, heart valve,...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Liver to muscle signal intensity ratio and T2* calculation versus liver iron concentration | during examination

SECONDARY OUTCOMES:
Difference between in-phase and out-phase T2* calculation versus liver fat concentration | during examination
Correlation between biochemical and MRI quantification of liver iron | during examination
Correlation between participating centers | during examination
Reproducibility of the multiecho gradient-echo sequence | during examination
Influence of the antenna for the multiecho gradient-echo sequence | during examination

CONTACTS AND LOCATIONS:
Overall Officials: Yves Gandon, MD, Study Director — Rennes University Hospital; Eric Bellissant, MD, PhD, Study Chair — Rennes University Hospital
Locations (10):
- France (9):
  - CHU Angers, Angers
  - Hôpital Beaujon, Clichy
  - Hôpital Huriez, Lille
  - Hôpital Edouard Herriot, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpital Saint Eloi, Montpellier
  - Hôpital Tenon, Paris
  - Hôpital de Pontchaillou, Rennes
  - Hôpital du Brabois, Vandœuvre-lès-Nancy
- Hopital Donostia-San Sebastian, Donostia / San Sebastian, Spain

REFERENCES:
- [Result] Paisant A, Boulic A, Bardou-Jacquet E, Bannier E, d'Assignies G, Laine F, Turlin B, Gandon Y. Assessment of liver iron overload by 3 T MRI. Abdom Radiol (NY). 2017 Jun;42(6):1713-1720. doi: 10.1007/s00261-017-1077-8. PMID 28224171
- [Result] Paisant A, Laine F, Gandon Y, Bardou-Jacquet E. Is room temperature susceptometer really an accurate method to assess hepatocellular iron? J Hepatol. 2017 Dec;67(6):1345-1346. doi: 10.1016/j.jhep.2017.07.021. Epub 2017 Aug 5. No abstract available. PMID 28789881
- [Result] d'Assignies G, Paisant A, Bardou-Jacquet E, Boulic A, Bannier E, Laine F, Ropert M, Morcet J, Saint-Jalmes H, Gandon Y. Non-invasive measurement of liver iron concentration using 3-Tesla magnetic resonance imaging: validation against biopsy. Eur Radiol. 2018 May;28(5):2022-2030. doi: 10.1007/s00330-017-5106-3. Epub 2017 Nov 24. PMID 29178028